CLINICAL TRIAL: NCT03600467
Title: A Single-arm, Open-label, Signal-seeking, Phase IIa Trial of the Activity of Seviteronel in Patients With Androgen Receptor (AR)-Positive GBM
Brief Title: Activity of Seviteronel in Patients With Androgen Receptor (AR)-Positive Glioblastoma
Acronym: START
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor
Sponsor: St Vincent's Hospital, Sydney (Other)
Responsible Party: Principal Investigator, Anthony Joshua, FRACP, Principle Investigator, St Vincent's Hospital, Sydney
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: START
Record Dates: First submitted 2018-06-22; First posted 2018-07-26 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Solid Tumor; Androgen Receptor Gene Overexpression
Keywords: Androgen Receptor Positive; Seviteronel; Advanced Cancers
MeSH Terms: interventions — seviteronel

STUDY DESIGN:
Intervention Model Description: START is an open-label, single-arm, multicentre Phase IIa signal-seeking trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adrogen Postive Solid Tumours (Experimental)
  Interventions: Drug: SEVI-D (Seviteronel in combination with dexamthasone)

INTERVENTIONS:
Drug: SEVI-D (Seviteronel in combination with dexamthasone) — Use of SEVI-D (Serivteronel and dexamethasone) in the treatment of androgen receptor positive solid tumours.
  Serivteronel will be administered orally at 450 mg (3 tables) once daily. It will be given in combination with one oral tablet of 0.5 mg tablet of Dexamethosone. SEVI-D will be continuously administered daily while on the study.
  Clinical and safety assessments are scheduled every 4 weeks during the study and then every 8 weeks after the end of the safety follow up period of the study.

SUMMARY:
This study's purpose is to facilitate and expedite the clinical testing of SEVI-D in a population with advanced GBM that are androgen receptor (AR) positive.

Who is it for? You may be eligible for this study if you have a GBM with clinical/radiological progression on or following last anticancer therapy.

Study details:

All participants will be screened to confirm if their GBM is AR positive by the study team. If eligible, participants will receive the medications of Serivteronel and Dexamethasone (also known as SEVI-D) by oral tablets continuously per cycle (4 weeks). Participants will be asked to have blood tests, scans, complete questionnaire and regularly meet with the study doctor and team.

It is hoped this research will demonstrate this treatment could be beneficial for the treatment of GBM that are known to be human androgen receptor positive.

DETAILED DESCRIPTION:
Background:

The human androgen receptor (AR) is a steroid hormone receptor that is expressed in multiple reproductive tissues and has important effects on multiple organ systems. The AR is a major target for the treatment of prostate cancer, and, more recently, for treatment of breast cancer. However, the AR is also expressed on many other tissues and plays vital roles in other cancer types, such as head and neck cancers (eg, salivary gland and thyroid cancers), cutaneous malignancies (eg, melanoma and basal cell carcinoma), sarcomas, and genitourinary cancers (eg, renal and bladder cancers). There are very few studies investigating AR-targeted therapies for indications other than prostate or breast cancer; however the few anecdotal reports and small studies that have been performed suggest that AR-positive tumours may respond to therapy with AR-targeted agents. In this study we are concentrating on GBM Seviteronel is a dual selective P450C17,20-lyase (CYP17 lyase) and AR inhibitor currently being investigated in Phase 1/2 trials for prostate and breast cancers. Seviteronel has shown promising preclinical activity in some breast cancer models, and seviteronel in combination with dexamethasone (SEVI-D) has shown promising preliminary activity for treatment of metastatic castration-resistant prostate cancer. Therefore, SEVI-D could be beneficial for the treatment of other cancers that are known to be AR-positive such as GBM

Aim:

The overall aim is to facilitate and expedite the clinical testing of rational therapeutic hypotheses in a population with advanced cancer and unmet need, with a particular, but not exclusive, focus on rare or neglected cancers. The program will evaluate the clinical activity of SEVI-D in subjects with AR-positive GBM

Primary Objective:

To test the clinical activity of novel targeted treatments and/or indications as measured by objective tumour response or the ratio of time-to-progression on study over the preceding period

Secondary Objectives:

1. Overall survival (OS) (death from any cause);
2. Safety and tolerability of treatment (rates of adverse events)
3. Health related quality of life during treatment (EORTC QLQ-C30v.3 questionnaire or brief pain inventory, if applicable).
4. To evaluate the feasibility, efficiency and utility of an overarching framework protocol for multiple, parallel signal-seeking clinical substudies;
5. To evaluate a mechanism for screening patients for actionable biomarkers to be used to guide therapy.

Population:

Patients with AR-positive GBM as confirmed by immunohistochemistry.

Treatments:

Seviteronel, will be administered orally at 450 mg (3 x 150 mg tablets) for men with 0.5 mg dexamethasone (tablet) once daily plus a GnRH analogue (depot injection). Seviteronel, will be administered orally at 450 mg (3 x 150 mg tablets) for post menopausal women, once daily in combination with once daily 0.5 mg dexamethasone (tablet). For premenopausal women (with intact ovaries), a GnRH analogue (depot injection) will also need to be admistered. See Treatment Study Table below. Patients will take seviteronel and dexamethasone each day continuously in 28-day cycles.

Assessments:

Screening for participation in the screening platform includes the review of patient history, current health status, availability of a biospecimen for AR screening and patient willingness to be in a trial if eligible.

Clinical and safety assessments are scheduled prior to registration and then every 8 weeks until death.

Imaging and other response assessments are required at baseline and 8-weekly from cycle 1 day 1 until progression.

Blood collection for translational studies will occur at:

1. Baseline (collected within 21 days prior to registration) or within 28 days of C1D1 treatment
2. Every 2nd cycle
3. At End of treatment

ELIGIBILITY:
Inclusion Criteria:

1. To be eligible for treatment in the study, patients must continue to meet all of the inclusion criteria and none of the exclusion criteria at the time of registration. Male or female patients, aged 18 years and older, with pathologically confirmed advanced GBM;
2. Sufficient and accessible tissue for molecular screening;
3. Patients receiving their last line of standard treatment or who have received and failed all standard anticancer therapy (where standard therapy exists) or have documented unsuitability for any further standard anticancer therapy Poor prognosis cancers or cancers with low expected response rate to standard treatment (in the opinion of the investigator and based on available evidence) may be screened on an earlier line of treatment.

   1. Failure is defined as either progression of disease (clinical or radiological) or intolerance to standard therapy resulting in the discontinuation of the therapy.
   2. Documented unsuitability for further standard therapy includes known hypersensitivity, organ dysfunction or other patient factors that would make therapy unsuitable in the judgement of the responsible investigator;
4. ECOG performance status 0, 1 or 2;
5. Willing and potentially able to comply with study requirements, including treatment, timing and/or nature of required assessments; It is the intention to screen patients who are in principle wishing to take part in the START study if they are found to have an appropriate tumour biomarker and are still eligible for enrolment at the time of the treatment phase;
6. Signed, written informed consent to participation in the molecular screening and treatment study.
7. Received and failed all standard anticancer therapy or have documented unsuitability for any further standard therapy, if standard therapy exists;
8. Clinical or radiological progression on or following last anticancer therapy;
9. Adequate organ system function as assessed by the following minimal laboratory requirements (within 7 days prior to first administration of study drug):

   1. bone marrow function; platelets ≥ 100 x 109/L, ANC ≥ 1.5 x 109/L, and haemoglobin ≥9g/dL (5.6mmol/L); white blood cell count ≥3,000 cells/μL
   2. liver function; ALT/AST ≤ 3 x ULN (in the absence of liver metastases, ≤ 5 x ULN for patients with liver involvement) and total bilirubin ≤1.5xULN;
   3. renal function; serum creatinine ≤1.5xULN;
10. Meet any additional inclusion criteria specified in the relevant study addendum;
11. Signed, written informed consent to participation in the specific treatment study.
12. AR-positive GBM confirmed by immunohistochemistry
13. Able to comply with study requirements

Exclusion Criteria:

Exclusion criteria will include those relevant for screening but also include:

1. Suitable for standard therapy or accepted standard care, if the patient has not been previously treated;
2. Specific comorbidities or conditions (e.g. psychiatric) or concomitant medications which may contraindicate participation and/or interact with seviteronel, dexamethasone or the GnRH analogue;
3. Other co-morbidities or conditions that may compromise assessment of key outcomes or in the opinion of the clinician, limit the ability of the patient to comply with the protocol;
4. For non central nervous system (CNS) cancers, patients with symptomatic CNS involvement of his/her cancer. Subjects with stable neurological function, on stable doses of steroids/anti-epileptics over 4 weeks, and with no evidence of CNS progression within 12 weeks prior to study entry are eligible;
5. History of another malignancy within 2 years prior to registration unless adequately treated and determined free of progressive and metastatic disease for at least 6 months. Patients with a past history of adequately treated carcinoma-in-situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or superficial transitional cell carcinoma of the bladder are eligible;
6. Pregnancy, lactation, or inadequate contraception. Women must be post-menopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration. Men must have been surgically sterilised or use a barrier method of contraception (double barrier, if required).
7. Known history of hypersensitivity to active or inactive components of seviteronel, dexamethasone, and/or GnRH analoge;
8. Previous treatment with seviteronel or same class of agent;
9. Treatment with any of the following anti-cancer therapies prior to the first dose of study treatment:

   * Radiation therapy, surgery or tumour embolization within 14 days prior to the first dose of study treatment. Palliative radiotherapy (for analgesia) is acceptable only if the irradiated field does not include target lesions;
   * Immunotherapy within 28 days prior to the first dose of study treatment;
   * Chemotherapy, biologic therapy, or hormonal therapy within 14 days or 5 half-lives of a drug prior to the first dose of study treatment or until recovery from previous therapy (whichever is longer);
10. Administration of any investigational treatment within 30 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study treatment;
11. Active prostate cancer requiring treatment.
12. Active breast cancer requiring treatment.
13. Symptomatic central nervous system cancer. Subjects with stable neurological function, on stable doses of steroids/anti-epileptics over 4 weeks prior to screening are eligible.
14. Corrected QT interval by the Fridericia correction formula (QTcF) on the screening electrocardiogram (ECG) >470 msec. If the screening ECG QTcF interval is >470 msec, it may be repeated once, and if the repeat ECG is <470 msec, the patient may be enrolled.
15. Clinically significant cardiac arrhythmias (eg, ventricular tachycardia, ventricular fibrillation, torsades de pointes, second degree or third degree atrioventricular heart block without a permanent pacemaker in place).
16. Any medical condition that could preclude patient participation in the study, pose an undue medical hazard, or which could interfere with study results.
17. Class III or IV Congestive Heart Failure as defined by the New York Heart Association functional classification system within the previous 6 months.
18. Known active Human Immunodeficiency Virus, Hepatitis B, or Hepatitis C infections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Objective tumour response or the ratio of time-to-progression over the preceding period | 1 year
  Assessing radiological images at each time point using either RECIST 1..1 or RANO criteria for disease progression.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  Number of Patients alive >= 5 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03. | Through study completion, average 1 year
  The type and frequency of treatment-related adverse events as assessed by CTCAE v4.03.
Change in quality of life measurements during treatment | Through study completion, average 1 year
  Change from Baseline in EORTC QLQ-C30 v3 questionnaires
Change in pain score measurements during treatment | Through study completion, average 1 year
  Change from Baseline in BP-SF questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- St Vincent's Hospital, Darlinghurst, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No